CLINICAL TRIAL: NCT07293117
Title: Evaluating Heart & Soil's Lifeblood on Iron and Energy Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 40434
Record Dates: First submitted 2025-12-05; First posted 2025-12-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Energy

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single Arm observational where participants act as their own control
  Interventions: Dietary Supplement: Heart & Soil Lifeblood

INTERVENTIONS:
Dietary Supplement: Heart & Soil Lifeblood — Lifeblood is an iron and blood-supporting supplement made of liver, spleen, and whole blood extract.

SUMMARY:
This study explores how Heart & Soil's Lifeblood impacts iron levels and energy.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to meticulously investigate the testimonials provided by individuals who have experienced changes in their iron levels and energy after using Heart & Soil's Lifeblood supplement. Recognizing the pivotal role of iron in red blood cell formation, oxygen transport, and numerous other physiological processes, this study aims to bridge the gap in current research concerning the effects of natural products, particularly freeze-dried organ extracts, on human biology. Unlike the extensively studied synthetic iron sulfate supplements, the study focuses on exploring the benefits of a natural alternative, aiming to enhance the understanding of how such products can support healthy iron stores and, by extension, improve overall vitality.

The objective of this study is to empower participants with personalized data and insights regarding their iron and energy levels. Through the evaluation of a comprehensive iron panel conducted before and after the supplementation of Lifeblood, investigators intend to establish a correlation between these iron levels and the perceptions of energy and fatigue, as reported through supplementary survey data. This approach transcends the realm of generic claims, delving into tangible, real-world outcomes that are directly influenced by participant engagement.

The specific aim is to quantify the impact of Lifeblood supplementation on iron levels and the subsequent enhancement of energy levels, thereby providing participants with personalized health insights. This will not only offer tailored feedback on how the supplement influences individual vitality but will also empower participants with the knowledge to make informed lifestyle decisions based on their unique health profiles.

The significance of this study lies in its potential to revolutionize the way individuals perceive and manage their energy levels through the consumption of natural, whole food, organ extracts. By integrating clinical studies with scientific rigor, investigators are set to validate the real-world experiences of individuals using supplementation to support their health. Although individual results may vary, the anticipated outcome is a personalized understanding of the role of iron in energy maintenance, presenting participants with a navigational tool for future wellness decisions. This study represents a pivotal step towards elevating our understanding of natural health products and their potential to enrich human health and vitality.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with Hemochromatosis
* Individuals with Severe Allergies
* Pregnant or Nursing Women
* Individuals with Gastrointestinal Disorders
* Individuals on Iron-Related Medications
* Individuals with Mental Health Disorders
* Competitive Athletes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-09 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Fatigue Perception and Impact Survey | Change from baseline (Day 1-7) in fatigue perception and impact at 4 to 5 weeks after the start of the intervention
  The Fatigue Perception and Impact Survey (FPIS) is a specialized questionnaire developed to evaluate the presence, severity, and impact of fatigue on an individual's life. Comprising a series of questions, the survey aims to capture both the subjective experience of fatigue and its consequences across various domains, such as physical, emotional, and social aspects. This tool is commonly used in clinical settings to assess fatigue in patients with various medical conditions, including chronic illnesses and cancer, helping healthcare professionals better understand and address the debilitating effects of fatigue on patients' quality of life. Researchers also employ the FPIS to gather valuable data on fatigue patterns, enabling a deeper understanding of the condition and potential interventions to alleviate its impact.
Iron and Ferritin Blood Levels | Change from baseline (Day 1-10) in iron and ferritin blood levels at 11 to 14 weeks after the start of the intervention
  Easily check your iron and ferritin levels at home with the MyLabsDirect test kit, featuring the Tasso specimen collection device. Simply clean your upper arm, apply the Tasso device, and press a button to painlessly collect a small blood sample in minutes. Secure your sample in the provided tube, package it, and mail it to MyLabsDirect's CLIA-certified lab for accurate results-no clinic visit required

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=40434